CLINICAL TRIAL: NCT01517867
Title: Comparing Two Parenting Programs for At-Risk Families
Brief Title: Early Parenting Intervention Comparison
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); University of Iowa (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00039328; R01NR012444 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Behavior Problems, Child
Keywords: preschool children behavior problems; child between 2 and 5 years old
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Chicago Parent Program arm (Experimental): The Chicago Parent Program is a 12-session group-based parenting skills training program
  Interventions: Behavioral: Chicago Parent Program
- Parent-Child Interaction Therapy (Active Comparator): Parent-Child Interaction Therapy is an individually tailored treatment for parents and children with behavior problems
  Interventions: Behavioral: Parent-Child Interaction Therapy

INTERVENTIONS:
Behavioral: Chicago Parent Program — The Chicago Parent Program is a 12-session group-based parenting skills intervention for parents of young children with behavior problems
  Arms: Intervention Chicago Parent Program arm
Behavioral: Parent-Child Interaction Therapy — Parent-Child Interaction Therapy is an individually-tailored coaching intervention for parents and young children with behavior problems
  Arms: Parent-Child Interaction Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of two parenting programs in a mental health clinic serving young children with behavior problems.

ELIGIBILITY:
Inclusion Criteria:

* child 2 to 5 years old
* parent reports reason for referral is child behavior problems
* parent is a biological or adoptive parent, or legal guardian of child

Exclusion Criteria:

* parent is psychotic or actively abusing substances
* child is autistic or severely developmentally delayed

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gross, DNSc, Principal Investigator — Johns Hopkins University, School of Nursing
Locations (1):
- The Family Center at Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing plan was developed.

REFERENCES:
- [Derived] Gross D, Belcher HME, Budhathoki C, Ofonedu ME, Dutrow D, Uveges MK, Slade E. Reducing Preschool Behavior Problems in an Urban Mental Health Clinic: A Pragmatic, Non-Inferiority Trial. J Am Acad Child Adolesc Psychiatry. 2019 Jun;58(6):572-581.e1. doi: 10.1016/j.jaac.2018.08.013. Epub 2018 Nov 12. PMID 30768419
- [Derived] Gross DA, Belcher HM, Ofonedu ME, Breitenstein S, Frick KD, Chakra B. Study protocol for a comparative effectiveness trial of two parent training programs in a fee-for-service mental health clinic: can we improve mental health services to low-income families? Trials. 2014 Mar 1;15:70. doi: 10.1186/1745-6215-15-70. PMID 24581245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Chicago Parent Program Arm | Parent-Child Interaction Therapy
Started | 81 | 80
Completed | 18 | 15
Not Completed | 63 | 65
Not completed — never started treatment | 29 | 32
Not completed — Withdrawal by Subject | 34 | 30
Not completed — Still in treatment at study end | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Chicago Parent Program Arm | Parent-Child Interaction Therapy | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Full Range); unit: years] | 33.0 [22 to 69] | 34.5 [22 to 71] | 33.76 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 75 | 148
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 76 | 78 | 154
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 59 | 114
  White | 16 | 18 | 34
  More than one race | 9 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Behavior Problems
Description: parent-report measure called The Child Behavior Checklist. Raw scores range from 0 to 198 with lower numbers being better for the child.
Time Frame: baseline, first follow-up (up to 2 years)
Population: First follow-up data collected from 42 participants in Chicago Parent Program and 34 participants in Parent-Child Interaction Therapy who started treatment and were discharged, regardless of whether they completed the full treatment. Did not collect follow-up data from remaining participants who enrolled in study but never attended any treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Chicago Parent Program Arm | Parent-Child Interaction Therapy
Number analyzed (Participants) | 42 | 34
units on a scale
  Baseline | 67.0 (13.42) | 67.6 (11.75)
  first follow-up (up to 2 years) | 60.4 (12.92) | 59.9 (13.34)

2. Secondary Outcome: Aggregate Cost
Description: Combined provider (based on billing records) and parent cost (based on self-report).
Time Frame: through end of study (up to 2 years)
Population: Cost collected for 42 participants in Chicago Parent Program and 34 participants in Parent-Child Interaction Therapy who started treatment and were discharged, regardless of whether they completed the full treatment. Did not collect cost data from the remaining participants who enrolled in study but never attended any treatment.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Intervention Chicago Parent Program Arm | Parent-Child Interaction Therapy
Number analyzed (Participants) | 42 | 34
dollars | 1413 (1211) | 2151 (2583)

ADVERSE EVENTS:
Time Frame: from the start of treatment until discharge (up to approximately 2 years)
Arm/Group | Intervention Chicago Parent Program Arm | Parent-Child Interaction Therapy
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 0/81 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT01517867/Prot_SAP_000.pdf